CLINICAL TRIAL: NCT01198925
Title: Assessment of the Optimal Dosing of Piperacillin-tazobactam in Intensive Care Unit Patients: Extended Versus Continuous Infusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/414
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Infectious Disease
Keywords: Infectious disease; piperacillin; continuous infusion; extended infusion
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- extended infusion (Active Comparator)
  Interventions: Drug: piperacillin extended infusion
- continuous infusion (Experimental)
  Interventions: Drug: piperacillin continuous infusion

INTERVENTIONS:
Drug: piperacillin continuous infusion — piperacillin continuous infusion
  Arms: continuous infusion
Drug: piperacillin extended infusion — piperacillin extended infusion
  Arms: extended infusion

SUMMARY:
Piperacillin-tazobactam is an acylureido-penicillin-beta-lactamase inhibitor combination and is frequently used in the empirical treatment of hospital-acquired infections because of its antipseudomonal activity. Similar to other beta-lactam antibiotics, piperacillin-tazobactam exhibits time-dependent killing and the T > MIC appears to be the best outcome predictor. Because a majority of infections are treated empirically, it is necessary to achieve a T > MIC equal to 50% of the dosing interval (50% T > MIC) against the most likely pathogens, including those with only moderate susceptibility The aim of this study is to compare the same dose of piperacillin/tazobactam administered by an extended infusion versus a continuous infusion. A pharmacokinetic study will be performed in patients treated by extended (loading dose 4 G/30 min followed by 4 X 4 G /3h) and continuous infusion (loading dose 4 G/30 min followed by 16G /24h).

A population pharmacokinetic analysis with Monte Carlo simulations will be used to determine 95% probability of target attainment (PTA95) versus MIC

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years) admitted on the intensive care unit (surgical and medical surgery).
* Starting a treatment with piperacillin/tazobactam
* Signed informed consent
* Hematocrit >= 21%
* Available arterial line

Exclusion Criteria:

* age <18 or >75 years
* patient's weight <50 or >100 kg
* renal insufficiency (estimated clearance < 50 ML /MIN)
* haemodialysis
* WBC < 1000 103 µl
* estimated survival <5 days
* meningitis or other proven infections of the CNS
* IgE-mediated allergy to penicillins
* pregnancy
* patients having participated in another study <30 days before inclusion in the present study
* retrospectively, marked deterioration of the renal function during the study period
* retrospectively, treatment < 96 h

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-09-23 (Actual); Primary Completion 2012-11-16 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics of piperacillin continuous infusion compared to piperacillin extended infusion | 6 hours
  Determination of serum concentrations of piperacillin.

SECONDARY OUTCOMES:
95% probability of target attainment (PTA95) versus MIC of different organisms. | 96 hours
  Determination of the probability of target attainment versus MIC of different organisms.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Decruyenaere, MD, PhD, Principal Investigator — University Hospital Ghent, Belgium
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website University Hospital Ghent, Belgium — http://www.uzgent.be